CLINICAL TRIAL: NCT06696365
Title: Intermittent Theta Burst Stimulation (iTBS) as a Treatment for Alcohol Use Disorder in Inpatient Treatment
Brief Title: iTBS for Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicholas Balderston, PhD (Other)
Responsible Party: Sponsor-Investigator, Nicholas Balderston, PhD, Assistant Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 856816
Record Dates: First submitted 2024-10-28; First posted 2024-11-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active iTBS (Experimental): The intermittent theta burst (iTBS) will be delivered using the MagVenture MagPro X100 stimulator equipped with a Cool B-70 A/P (combined active & sham) figure of eight coil. Treatment will be at 100% of MT. Treatment will be approximately 2 ½ minutes long. Each session will be 2-hours in length and consist of four treatments spaced 30 minutes apart. There will be a total of five sessions over the course of five to seven days.
  Interventions: Device: TMS
- Sham iTBS (Sham Comparator): The B70 A/P coil is also equipped with an active sham electric stimulation (e-stim) system that delivers a small current pulse synchronous to the TMS pulse, titrated to match the TMS sensations. This pulse is similar in duration and distribution to the current induced by the TMS pulse . This pulse will be delivered to the scalp adjacent to the stimulation site via disposable low-profile webbed EEG electrodes filled with electrolytic gel. Electrodes will be connected to the e-stim system via one of two identical cables allowing the operator to deliver either real or sham electric stimulation. Cables will be labeled to match the corresponding coil side so that each session always includes either active TMS or active e-stim, but never both.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The intermittent theta burst (iTBS) will be delivered using the MagVenture MagPro X100 stimulator equipped with a Cool B-70 A/P (combined active & sham) figure of eight coil. MagVenture MagPro X100 is available commercially and has been FDA approved to treat major depressive disorder and obsessive-compulsive disorder.

SUMMARY:
The two primary objectives of this study are to test whether intermittent theta-burst (iTBS) can affect behavioral change as compared to treatment as usual (TAU, sham) in individuals with alcohol use disorder (AUD) in inpatient substance use treatment. The secondary objective is to determine whether iTBS reduces the risk for relapse at four months compared to sham. It is hypothesized that individuals who receive iTBS treatment will show attenuated prefrontal cortex (PFC) CNS responses to alcohol related cues and reductions in risk-taking behavior and impulsivity as measured by PFC responses measured by functional near infrared spectroscopy (fNIRs). The proposed approach will be to measure the effect of iTBS treatment on PFC CNS response. Participants will be randomized to receive 5 days (4 x sessions/day x 600 pulses/session = 12,000 pulses) of iTBS or sham to the left dorsal lateral prefrontal cortex (dlPFC) while being exposed to alcohol cues five minutes prior to treatment and during treatment. The investigators will target the Beam/F3 scalp location and use the TMS Navigator Research Premium stereotaxic system for neuronavigation. PFC response data will be gathered using fNIRs measuring cue reactivity, risk-taking (Balloon Analog Risk Test), and impulsiveness (Go No Go task). The primary outcomes will be the mean changes in pre-post PFC response data gathered using the fNIRs sessions. The rationale for this approach is that TBS can be delivered over a shorter time frame than rTMS and may require fewer sessions, allowing for a better fit within a 28-day inpatient treatment stay.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged >21and <75
4. Right-handed
5. Diagnosed with an AUD disorder seeking treatment at Caron Treatment Centers and planning to be enrolled in residential treatment for a minimum of 28 days.
6. Ability to obtain an MT at the first session.
7. Women of childbearing potential must consent to use a medically accepted method of birth control (e.g., implants, injectables, oral contraceptives, IUD, sexual abstinence, or vasectomized partner) or to abstain from sexual intercourse only during the five treatment days of the study.

Exclusion Criteria:

1. Age <21 or >75 years.
2. Women who are pregnant, planning pregnancy, breastfeeding, or unwilling to use adequate contraceptive measures.
3. Evidence or history of a significant neurological disorder including moderate-severe head trauma, stroke, Parkinson's disease, or other movement disorder (except benign essential tremor), epilepsy. History of seizures (except juvenile febrile seizures or any condition/concurrent medication that could notably lower seizure threshold. This may include traumatic brain injury (TBI) if the TBI places the individual at an elevated risk of seizure.
4. Have a cardiac pacemaker.
5. Have an implanted device or metal in the brain.
6. Have a cochlear implant.
7. Have a current amnestic disorder, delirium, or other cognitive disorder.
8. Previous treatment with TMS.
9. Left-handed
10. Suicidal ideation within the past month, or history of suicide attempt(s) within the past year.
11. Active psychosis or history of severe psychiatric disorder with psychosis or unstable or untreated psychiatric disorder with potential for psychosis.
12. Abnormal physical exam findings, vital signs (blood pressure, heart rate, respiratory rate, body temperature), EKG measurements, and safety lab values that are deemed clinically significant by a study physician.
13. Diagnoses of severe depression or bipolar disorder.
14. Anyone who in the opinion of the principal investigator (PI) or study physician would not be appropriate for participation (i.e., behavioral issues during clinical treatment, clinical needs outweighing research participation).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Cue-evoked prefrontal cortex activity | 24 hours before first iTBS session and 24 hours after last iTBS session
  Individuals will undergo a cue reactivity task composed of four stimulus categories: general alcohol cues; alcohol cues specific to patient alcohol choice preferences; natural reward cues; and emotionally neutral cues (e.g., pictures of everyday objects like lamps, pens) will be monitored with Functional near-infrared spectroscopy (fNIRS) over the prefrontal cortex. fNIRS measures the amount of infrared light absorbed by the brain, which differs as a function of ongoing brain activity. The magnitude of this signal (absorption factor) will be calculated for the conditions described above.

SECONDARY OUTCOMES:
Risk-taking | 24 hours before first iTBS session and 24 hours after last iTBS session
  The Balloon Analog Risk Task (BART) will be used to measure risk-taking behavior. Participants are presented with virtual balloons that they must blow up, but not pop. The more they fill their virtual balloons, the greater the reward. However, if the balloon pops, they lose their rewards. The primary measure of this task it the average number of pumps per balloon, which is a measure of their risk-taking behavior.
Impulsiveness | 24 hours before first iTBS session and 24 hours after last iTBS session
  The Go/No Go task will be used to measure impulsiveness. Participants are given a series of trials where they are required to respond to the go stimuli and withhold a response to the no-go stimuli. Performance on this task will be assessed by comparing their accuracy on the go trials to their accuracy on the no-go trials using d-prime (Hits - False alarms), which is associated with impulsive responding on the no-go trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Caron Treatment Centers, Wernersville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No